CLINICAL TRIAL: NCT04344873
Title: Impact of T Cells on Age-related Vascular Dysfunction: A Translational Approach
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID initially delayed plans to begin recruitment of subjects. Subsequently, the departure of a clinical investigator and loss of access to equipment and study subject population resulted in study termination before any subjects were enrolled.
Sponsor: University of Utah (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Anthony (Tony) Donato, Associate Professor, Geriatrics, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB_00118392; R01AG060395 (NIH)
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Inflammation; Aging
Keywords: Aging; Inflammation; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: Prospective placebo controlled crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Older Adult participants (Experimental): Older adult participants (ages 55-75) will be assessed for arterial function using FMD analysis, PWV calculations, T Cell phenotyping, and proportion of inflammatory biomarkers after injections of placebo and abatacept.
  Interventions: Other: Placebo; Drug: Abatacept 10 mg/kg

INTERVENTIONS:
Other: Placebo — Placebo injection at day one and day fourteen.
Drug: Abatacept 10 mg/kg — Abatacept injection at day twenty eight and day forty two.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in the United States and other industrialized societies, and advanced age is the major risk factor for development of CVD. Advancing age appears to exert its pathological influence primarily via adverse functional and structural effects on arteries. Aging is associated with increased stiffness (reduced compliance) of large elastic arteries and impaired arterial endothelial function that is characterized by reductions in nitric oxide (NO)- mediated endothelium-dependent dilation (EDD). While several changes to arteries may contribute to age-associated increases in CVD risk; the development of endothelial dysfunction and stiffening of the large elastic arteries are among the most important contributors. Both are predictors of CV events and clinical CVD with increasing age. Although the importance of endothelial dysfunction and arterial stiffening with age are well established, the initiating events of these deleterious changes are elusive.

DETAILED DESCRIPTION:
Advanced age is the primary and most predictive risk factor for CVD. The investigators have demonstrated that there is a pronounced age-associated increase in T cell infiltration into the perivascular space around large elastic arteries and small resistance arteries. The objective of this study is to determine if and how T cells contribute to age-related arterial inflammation and dysfunction.

Although there is evidence from rodent studies that T cells play a critical role in arterial dysfunction, it is unknown whether this occurs in humans. Abatacept, a T cell co-stimulation inhibitor, is FDA approved for treatment of rheumatoid arthritis. Importantly, Abatacept decreases the inflammatory phenotype of circulating T cells. Abatacept will be used in older adults to be the first to determine if T cell inflammation contributes to arterial dysfunction in older adults. The investigators hypothesize that older adults treated with Abatacept will exhibit greater flow-mediated dilation, decreased pulse wave velocity, decreased or unchanged blood pressure, decreased inflammatory and oxidative stress markers in endothelial cells, decreased plasma free radicals, decreased proportion of memory T cells, and experience a shift away from a pro-inflammatory T cell phenotype compared to placebo. These results will be interpreted to mean that T cells play a role in mediating age-related arterial dysfunction in humans.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (55-75 years old).
* Women will be at least two years postmenopausal, not using hormone therapy and have a follicle stimulating hormone (FSH) concentration of >30 IU/L.

Exclusion Criteria:

* Autoimmune disorders,
* Hypertension (blood pressure >140/90mmHg),
* Body mass index of >30 kg/m2,
* Clinical CVD,
* Diabetes
* Current tobacco use,
* Regular aerobic exercise (>30 mins per day, > 2 days per week for the at least the last 2 years),
* Current or recurring infections within 12 weeks of the baseline visit,
* A positive tuberculosis (TB) test or subjects at risk of TB,
* Positive test for Hepatitis B, C, or cytomegalovirus (CMV),
* Use of immunosuppressive medication,
* Vaccination within 4 weeks of the baseline visit,
* Major surgery within 8 weeks of the baseline visit,
* Previous lymphoid irradiation or bone marrow transplant,
* Subjects at risk for diverticulitis,
* Any laboratory test result that, in the opinion of the overseeing physician (Dr. Frech) might place a participant at unacceptable risk.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in brachial arterial diameter after abatacept injection. | 7 weeks
Change in brachial arterial flow rate after abatacept injection. | 7 weeks

SECONDARY OUTCOMES:
Change in pulse wave velocity as measured by doppler ultrasound after abatacept injection. | 7 weeks
Change in proportion of memory T-Cells after abatacept injection | 7 weeks
Change in proportion of inflammatory biomarker Tumour Necrosis Factor alpha (TNF-α) after abatacept injection | 7 weeks
Change in proportion of inflammatory biomarker Interferon gamma (IFN-γ) after abatacept injection | 7 weeks
Change in proportion of inflammatory biomarker interleukin 10 (IL-10) after abatacept injection | 7 weeks
Change in proportion of inflammatory biomarker interleukin 17 (IL-17) after abatacept injection | 7 weeks
Change in proportion of inflammatory biomarker forkhead box P3 (FoxP3) after abatacept injection | 7 weeks
Change in proportion of inflammatory biomarker perforin after abatacept injection | 7 weeks

IPD SHARING:
Plan to Share IPD: No